CLINICAL TRIAL: NCT03428022
Title: Apatinib Combined With Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors Used for the Advanced Slow-progressed Non Small Cell Lung Cancer Patients With EGFR-TKI Resistance
Brief Title: Apatinib Combined With EGFR-TKI for Advanced Slow-progressed EGFR-TKI Resistant NSCLC
Acronym: AFLC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen People's Hospital (Other)
Responsible Party: Principal Investigator, Cao，Hua, associate chief physician, Shenzhen People's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFLC
Record Dates: First submitted 2018-01-15; First posted 2018-02-09 (Actual); Last update posted 2019-04-04 (Actual); Status verified 2019-04

CONDITIONS: NSCLC; Apatinib; EGFR-TKI
Keywords: Apatinib; EGFR-TKI resistance; slowly progress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Apatinib combined with EGFR-TKI (Experimental): Apatinib（Tablet（Tab. ）500millgram（mg）/day（d）） combined with EGFR-TKI（as previously）
  Interventions: Drug: Apatinib（Tab. 500mg/d） combined with EGFR-TKI（as previously）

INTERVENTIONS:
Drug: Apatinib（Tab. 500mg/d） combined with EGFR-TKI（as previously） — Patients with advanced non-small cell lung cancer (NSCLC) who had treated with EGFR-TKI and progressed slowly because of resistance are underwent with apatinib mesylate and continuous EGFR-TKI.

SUMMARY:
Patients with advanced non-small cell lung cancer (NSCLC) who progress slowly after Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors（EGFR-TKI）resistance will be treated with Apatinib and EGFR-TKI. The primary objective is the disease progression free survival of the patients.

DETAILED DESCRIPTION:
Patients with advanced non-small cell lung cancer (NSCLC) who had treated with Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors（EGFR-TKI） and progressed slowly because of resistance are underwent with apatinib mesylate and continuous EGFR-TKI. The primary objective is the disease progression free survival of the patients. The secondary goals are overall survival, duration of response, objective response rates, disease control rates, quality of life scores and drug safety. Currently such patients are treated with EGFR-TKI continuously, but 3 months later, the disease will be progressed rapidly. This study will bring a new treatment that are more effective, less toxic and more convenient for NSCLC-patients with EGFR-TKI resistance.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically confirmed advanced (stage IV) non-squamous, non-small cell lung cancer with measurable lesions
* Electronics Coordinating Grop（ECOG）score：0-2
* Expected survival over 3months
* Hemoglobin(HB)≥90 gram(g)/liter(L)；absolute neutrophil count(ANC)≥1.5×109/L；platelet(PLT)≥80×109/L；total-bilirubin（T-BIL）<1.5 upper limit of normal value（ULN）；alanine aminotransferase（ALT）and aspartate aminotransferase（AST）<2.5 ULN；Cr≤1.25ULN

Exclusion Criteria:

* Brain metastases, meningococcal meningitis, patients with spinal cord compression with evidence of imaging (computed tomography（CT） / magnetic resonance imaging （MRI）, et cetera（etc.）);
* Uncontrolled hypertension (systolic blood pressure（BP）≥140 millimeter mercury column（mmHg） or diastolic BP ≥90 mmHg, despite optimal drug therapy);
* Hemorrhoid dysfunction (inernational standard ratio(INR)> 1.5 or prothrombin time (PT)> ULN + 4 seconds or activated partial thromboplastin(APTT)> 1.5 ULN) with bleeding tendency or undergoing thrombolytic or anticoagulant therapy;
* Patients treated with anticoagulants or vitamin K antagonists such as warfarin, heparin, or the like;
* Patients underwent major surgery or severe traumatic injury, fracture or ulcer in 4 weeks before study;
* Urine routine urine protein ≥ +++, or confirmed 24 hours urinary protein content ≥ 1.0 g;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2017-12-01 (Actual); Primary Completion 2020-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | 3 months
  the disease progression free survival of patients

SECONDARY OUTCOMES:
OS | 8 months
  overall survival
ORR | 6 months
  objective response rates

CONTACTS AND LOCATIONS:
Overall Officials: CAO HUA, MD, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China